CLINICAL TRIAL: NCT01764841
Title: Randomized, Double-blind, Placebo-controlled, Multicenter Study Comparing Ciprofloxacin DPI 32.5 mg BID (Twice a Day) Intermittently Administered for 28 Days on / 28 Days Off or 14 Days on / 14 Days Off Versus Placebo to Evaluate the Time to First Pulmonary Exacerbation and Frequency of Exacerbations in Subjects With Non-Cystic Fibrosis Bronchiectasis.
Brief Title: Ciprofloxacin Dry Powder for Inhalation in Non-cystic Fibrosis Bronchiectasis (Non-CF BE)
Acronym: RESPIRE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15625; 2011-004208-39 (EudraCT Number)
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Bronchiectasis
Keywords: Ciprofloxacin; Dry Powder for Inhalation; Exacerbation; Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ciprofloxacin DPI 28 Days on/off (Cipro 28) (Experimental): Participants received ciprofloxacin (BAYQ3939) 32.5 milligram (mg) corresponding to 50 mg dry powder for inhalation (DPI) administered twice daily (BID) (every 12 hours); a treatment cycle consisted of a 28-day on-treatment phase followed by a 28-day off-treatment phase (48 weeks treatment phase = 6 active cycles).
  Interventions: Drug: Ciprofloxacin DPI (BAYQ3939)
- Ciprofloxacin DPI 14 Days on/off (Cipro 14) (Experimental): Participants received ciprofloxacin 32.5 mg corresponding to 50 mg DPI administered BID (every 12 hours); a treatment cycle consisted of a 14-day on-treatment phase followed by a 14-day off-treatment phase (48 weeks treatment phase = 12 active cycles).
  Interventions: Drug: Ciprofloxacin DPI (BAYQ3939)
- Placebo 28 Days on/off (Placebo 28) (Placebo Comparator): Participants received placebo matched to ciprofloxacin 32.5 mg powder (containing 40 mg dry powder) administered BID (every 12 hours); a treatment cycle consisted of a 28-day on-treatment phase followed by a 28-day off-treatment phase (48 weeks treatment phase = 6 cycles).
  Interventions: Drug: Placebo
- Placebo 14 Days on/off (Placebo 14) (Placebo Comparator): Participants received placebo matched to ciprofloxacin 32.5 mg powder (containing 40 mg dry powder) administered BID (every 12 hours); a treatment cycle consisted of a 14-day on-treatment phase followed by a 14-day off-treatment phase (48 weeks treatment phase = 12 cycles).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin DPI (BAYQ3939) — Participants received 32.5 mg ciprofloxacin hydrated (corresponding to 50 mg dry powder) administered BID (every 12 hours) using T-326 powder inhaler device.
  Arms: Ciprofloxacin DPI 14 Days on/off (Cipro 14); Ciprofloxacin DPI 28 Days on/off (Cipro 28)
Drug: Placebo — Participants received placebo matched to ciprofloxacin 32.5 mg powder (containing 40 mg dry powder) administered BID (every 12 hours) using T-326 powder inhaler device.
  Arms: Placebo 14 Days on/off (Placebo 14); Placebo 28 Days on/off (Placebo 28)

SUMMARY:
The purpose of this study is to evaluate if the time to first pulmonary exacerbation of bronchiectasis or its frequency can be prolonged by inhalation of ciprofloxacin for 28 days every other 28 days or for 14 days every other 14 days over 48 weeks.

DETAILED DESCRIPTION:
Number of participants with Adverse events will be covered in Adverse Events section.

The statistical analysis tests for the efficacy variables will be performed hierarchically. The comparisons ciprofloxacin DPI vs. pooled placebo (according to statistical analysis plan defined for FDA registration) will be performed in parallel for the regimen 28 days on/off and 14 days on/off.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a proven and documented diagnosis of non Cystic Fibrosis (CF) idiopathic or post infectious bronchiectasis
* Stable pulmonary status and stable regimen of standard treatment at least for the past 4 weeks

Exclusion Criteria:

* Forced expiratory volume in 1 second (FEV1) <30% or >90% predicted
* Active allergic bronchopulmonary aspergillosis
* Active and actively treated non tuberculosis mycobacterial (NTM) infection or tuberculosis
* Primary diagnosis of Chronic obstructive pulmonary disease (COPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2013-05-02 (Actual); Primary Completion 2016-03-09 (Actual); Study Completion 2016-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (135):
- United States (37):
  - Jasper, Alabama
  - Flagstaff, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Fort Smith, Arkansas
  - Los Angeles, California
  - Torrance, California
  - Ventura, California
  - Farmington, Connecticut
  - Waterbury, Connecticut
  - Washington D.C., District of Columbia
  - Celebration, Florida
  - Miami, Florida
  - Orlando, Florida
  - Weston, Florida
  - Winter Park, Florida
  - Lawrenceville, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Michigan City, Indiana
  - Hazard, Kentucky
  - Chesterfield, Missouri
  - Summit, New Jersey
  - New Hyde Park, New York
  - New York, New York
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Fort Worth, Texas
  - Houston, Texas
  - Kingwood, Texas
  - McKinney, Texas
  - Tyler, Texas
  - Abingdon, Virginia
  - Richmond, Virginia
  - Spokane, Washington
  - Tacoma, Washington
- Argentina (3):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Godoy Cruz, Mendoza Province
  - Vicente López
- Australia (11):
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Woodville, South Australia
  - Parkville, Victoria
  - Prahran, Victoria
  - Murdoch, Western Australia
  - Box Hill
  - Cairns
  - Frankston
  - Kogarah
  - Toorak Gardens
- Denmark (4):
  - Aarhus C
  - Hellerup
  - Næstved
  - Roskilde
- France (4):
  - Clermont-Ferrand
  - Montpellier
  - Nîmes
  - Toulon
- Germany (10):
  - Heidelberg, Baden-Wurttemberg
  - Cottbus, Brandenburg
  - Frankfurt am Main, Hesse
  - Neu-Isenburg, Hesse
  - Hanover, Lower Saxony
  - Koblenz, Rhineland-Palatinate
  - Geesthacht, Schleswig-Holstein
  - Jena, Thuringia
  - Berlin
  - Hamburg
- Israel (9):
  - Afula
  - Ashkelon
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- Italy (10):
  - Bari, Apulia
  - Benevento, Campania
  - Trieste, Friuli Venezia Giulia
  - Rome, Lazio
  - Pavia, Lombardy
  - Varese, Lombardy
  - Cagliari, Sardinia
  - Catania, Sicily
  - Pisa, Tuscany
  - Verona, Veneto
- Japan (10):
  - Tōon, Ehime
  - Nakagun, Ibaraki
  - Kōshi, Kumamoto
  - Matsusaka, Mie-ken
  - Tsu, Mie-ken
  - Sakai, Osaka
  - Hamamatsu, Shizuoka
  - Kiyose, Tokyo
  - Mitaka, Tokyo
  - Fukuoka
- Latvia (5):
  - Daugavpils
  - Jūrmala
  - Krāslava
  - Riga
  - Talsu
- New Zealand (6):
  - Auckland
  - Christchurch
  - Dunedin
  - Hamilton
  - Tauranga
  - Wellington
- Slovakia (2):
  - Bratislava
  - Prešov
- Spain (13):
  - Santiago de Compostela, A Coruña
  - Elda, Alicante
  - Badalona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Sant Boi de Llobregat, Barcelona
  - Terrassa, Barcelona
  - Pozuelo de Alarcón, Madrid
  - Oviedo, Principality of Asturias
  - Barcelona
  - Cáceres
  - Madrid
  - Pontevedra
  - Valencia
- United Kingdom (11):
  - Cambridge, Cambridgeshire
  - Exeter, Devon
  - Plymouth, Devon
  - Torbay, Devon
  - Dundee, Dundee City
  - Belfast, North Ireland
  - Shrewsbury, Shropshire
  - Newcastle upon Tyne, Tyne and Wear
  - London
  - Londonderry
  - Manchester

REFERENCES:
- [Derived] De Soyza A, Aksamit T, Bandel TJ, Criollo M, Elborn JS, Operschall E, Polverino E, Roth K, Winthrop KL, Wilson R. RESPIRE 1: a phase III placebo-controlled randomised trial of ciprofloxacin dry powder for inhalation in non-cystic fibrosis bronchiectasis. Eur Respir J. 2018 Jan 25;51(1):1702052. doi: 10.1183/13993003.02052-2017. Print 2018 Jan. PMID 29371383
- [Derived] Aksamit T, Bandel TJ, Criollo M, De Soyza A, Elborn JS, Operschall E, Polverino E, Roth K, Winthrop KL, Wilson R. The RESPIRE trials: Two phase III, randomized, multicentre, placebo-controlled trials of Ciprofloxacin Dry Powder for Inhalation (Ciprofloxacin DPI) in non-cystic fibrosis bronchiectasis. Contemp Clin Trials. 2017 Jul;58:78-85. doi: 10.1016/j.cct.2017.05.007. Epub 2017 May 8. PMID 28495619
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 124 study centers in 14 countries (Argentina, Australia, Denmark, France, Germany, Israel, Italy, Japan, Latvia, New Zealand, Slovakia, Spain, UK and US) between 02 May 2013 (first subject first visit) and 09 March 2016 (last subject last visit).
Pre-assignment Details: Overall 902 participants were screened, of them 486 were screen failures, and 416 were randomized, out of which 414 participants were assigned to the treatment. One participant from Ciprofloxacin 14 Days on/off group and one participant from Placebo 28 Days on/off group did not receive the study treatment after initial screening.
Period: Overall Study
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Placebo 28 Days on/Off (Placebo 28) | Placebo 14 Days on/Off (Placebo 14)
Started | 141 | 137 | 70 | 68
Participants Received Treatment | 141 (safety population) | 136 (safety population) | 69 (safety population) | 68 (safety population)
Completed | 118 | 111 | 56 | 49
Not Completed | 23 | 26 | 14 | 19
Not completed — Logistical Difficulties | 0 | 1 | 0 | 0
Not completed — Death | 3 | 0 | 1 | 4
Not completed — No Follow Up | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 24 | 11 | 15
Not completed — Lost to Follow-up | 3 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Placebo 28 Days on/Off (Placebo 28) | Placebo 14 Days on/Off (Placebo 14) | Total
Number analyzed (Participants) | 141 | 137 | 70 | 68 | 416
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (12.1) | 65.2 (13.5) | 64 (13.5) | 65.5 (12.9) | 64.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 88 | 52 | 44 | 285
  Male | 40 | 49 | 18 | 24 | 131
Saint George's Respiratory Questionnaire (SGRQ) Symptoms Component Score [Mean (Standard Deviation); unit: Score on a scale] — The SGRQ was a validated, disease-specific instrument that measures health-related quality of life (HRQoL) in adults with chronic obstructive pulmonary disease (COPD) and asthma and was later validated for use in bronchiectasis. The SGRQ covers 3 dimensions: symptoms, activity and impact on daily life. To determine the outcome, a score ranging from 1 to 100 was calculated for each individual domain and for the total score, and smaller scores indicate better health status. For this baseline measure, the symptoms component score was reported. Population: Participants with data available for this measure at baseline.
  Score on a scale
    number analyzed (Participants) | 135 | 129 | 67 | 66 | 397
    (all) | 60.72 (19.47) | 52.51 (21.48) | 55.52 (22.07) | 58.72 (20.4) | 56.84 (20.95)
Quality of Life Questionnaire for Bronchiectasis (QoL-B) Respiratory Symptoms Domain Score [Mean (Standard Deviation); unit: Score on a scale] — The QoL-B was a disease-specific questionnaire developed for non-Cystic fibrosis Bronchiectasis. It covers 8 dimensions: physical functioning, role functioning, emotional functioning, social functioning, vitality, treatment burden, health perceptions, and respiratory symptoms. Each dimension was scored separately on a scale of 0 to 100, and higher scores represent better outcomes. For this baseline measure, the respiratory symptoms domain score was reported. Population: Participants with data available for this measure at baseline.
  Score on a scale
    number analyzed (Participants) | 128 | 120 | 63 | 65 | 376
    (all) | 53.01 (18.71) | 57.69 (18.72) | 55.82 (18.04) | 50.67 (19.59) | 54.57 (18.87)
Forced Expiratory Volume in One Second (FEV1) [Mean (Standard Deviation); unit: Liter] — FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration, expressed in liters at body temperature and ambient pressure saturated with water vapor (BTPS).
  Liter | 1.521 (0.521) | 1.528 (0.625) | 1.577 (0.651) | 1.468 (0.574) | 1.524 (0.587)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Exacerbation Event Within 48 Weeks
Description: Time to first exacerbation was defined as the time from randomization until the visit at which the first qualifying exacerbation is recorded by the investigator. Exacerbation events are defined as exacerbations with systemic antibiotic use and presence of fever or malaise / fatigue and worsening of at least three signs/symptoms.
Time Frame: Up to Week 48
Population: Full analysis set (FAS) included participants who were randomized.
Measure: Median (97.5% Confidence Interval); unit: Days
Groups:
- Pooled Placebo: Participants received placebo matched to ciprofloxacin 32.5 mg powder (containing 40 mg dry powder) administered BID (every 12 hours); a treatment cycle consisted of a 28-day or 14-day on-treatment phase followed by a 28-day or 14-day off-treatment phase (48 weeks treatment phase = 6 or 12 cycles).
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Number analyzed (Participants) | 141 | 137 | 138
Days | 336 [206 to NA] — Value cannot be estimated due to censored data. | NA [290 to NA] — Value cannot be estimated due to censored data. | 186 [136 to 282]
Statistical Analysis 1: Comparison: Ciprofloxacin DPI 28 Days on/Off (Cipro 28) vs Pooled Placebo; The hazard ratio for time to first exacerbation event within 48 weeks and 97.5% Confidence Interval (CI) was calculated by using Cox proportional hazards model by comparison of Cipro 28/Pooled Placebo reporting groups. P-value was analysed using Wald-type test; Test type: Superiority or Other; p = 0.0650, Wald-type test; Hazard Ratio (HR) = 0.7331, 97.5% CI 2-sided [0.5027 to 1.0690]
Statistical Analysis 2: Comparison: Ciprofloxacin DPI 14 Days on/Off (Cipro 14) vs Pooled Placebo; The hazard ratio for time to first exacerbation event within 48 weeks and 97.5% CI was calculated by using Cox proportional hazards model by comparison of Cipro 14/Pooled Placebo reporting groups. P-value was analysed using Wald-type test; Test type: Superiority or Other; p = 0.0005, Wald-type test; Hazard Ratio (HR) = 0.5333, 97.5% CI 2-sided [0.3568 to 0.7971]

2. Secondary Outcome: Number of Participants With Exacerbation Events With Worsening of at Least Three Signs/Symptoms Over 48 Weeks
Description: For this outcome measure, exacerbation events were defined as exacerbations with systemic antibiotic use and presence of fever or malaise / fatigue and worsening of at least three signs/symptoms over 48 weeks.
Time Frame: Up to Week 48
Population: Full analysis set (FAS) included participants who were randomized.
Measure: Number; unit: Participants
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Number analyzed (Participants) | 141 | 137 | 138
Participants
  Number of exacerbations: 0 | 66 | 72 | 44
  Number of exacerbations: 1 | 44 | 38 | 58
  Number of exacerbations: 2 | 12 | 13 | 19
  Number of exacerbations: 3 | 12 | 8 | 7
  Number of exacerbations: 4 | 3 | 3 | 8
  Number of exacerbations: 5 | 1 | 2 | 0
  Number of exacerbations: 6 | 0 | 0 | 1
  Number of exacerbations: 7 | 3 | 1 | 1
Statistical Analysis 1: Comparison: Ciprofloxacin DPI 28 Days on/Off (Cipro 28) vs Pooled Placebo; A Poisson regression with adjustment for over-/under dispersion was used to analyze the number of exacerbation events over 48 weeks and to test the difference in the frequency of exacerbation between Ciprofloxacin DPI 28 and Pooled placebo group. P-value was analyzed using Wald-type test along with the incidence rate ratio of the comparison; Test type: Superiority or Other; p = 0.2944, Poisson regression; Incidence Rate Ratio = 0.8615, 97.5% CI 2-sided [0.6264 to 1.1848]
Statistical Analysis 2: Comparison: Ciprofloxacin DPI 14 Days on/Off (Cipro 14) vs Pooled Placebo; A Poisson regression with adjustment for over-/under dispersion was used to analyze the number of exacerbation events over 48 weeks and to test the difference in the frequency of exacerbation between Ciprofloxacin DPI 14 and Pooled placebo group. P-value was analyzed using Wald-type test along with the incidence rate ratio of the comparison; Test type: Superiority or Other; p = 0.0382, Poisson regression; Incidence Rate Ratio = 0.7329, 97.5% CI 2-sided [0.5237 to 1.0256]

3. Secondary Outcome: Number of Participants With Exacerbation Events With Worsening of at Least One Sign/Symptom Over 48 Weeks
Description: For this outcome measure, exacerbation events were defined as exacerbations with systemic antibiotic use and worsening of at least one sign/symptom over 48 weeks.
Time Frame: Up to Week 48
Population: Full analysis set (FAS) included participants who were randomized.
Measure: Number; unit: Participants
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Number analyzed (Participants) | 141 | 137 | 138
Participants
  Number of exacerbations: 0 | 58 | 68 | 46
  Number of exacerbations: 1 | 47 | 42 | 43
  Number of exacerbations: 2 | 12 | 15 | 31
  Number of exacerbations: 3 | 14 | 5 | 11
  Number of exacerbations: 4 | 4 | 2 | 5
  Number of exacerbations: 5 | 4 | 3 | 2
  Number of exacerbations: 6 | 2 | 2 | 0

4. Secondary Outcome: Percentage of Participants With Pathogen Eradication at End of Treatment (Week 44/46)
Description: Pathogen eradication was defined as a negative culture result for all pre-specified pathogens at end of treatment (week 44 or 46 depending on treatment regimen) that were present in the participant at baseline. There was no imputation for participants who discontinued the study prematurely.
Time Frame: End of treatment (Week 44/46)
Population: Full analysis set (FAS) included participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Number analyzed (Participants) | 141 | 137 | 138
Percentage of Participants
  No | 39.0 | 26.3 | 33.3
  Yes | 24.1 | 28.5 | 16.7

5. Secondary Outcome: Mean Change From Baseline in Patient Reported Outcome Saint George's Respiratory Questionnaire (SGRQ) Symptoms Component Score at End of Treatment (Week 44/46)
Description: The SGRQ was a validated, disease-specific instrument that measures health-related quality of life (HRQoL) in adults with chronic obstructive pulmonary disease (COPD) and asthma and was later validated for use in bronchiectasis. The SGRQ covers 3 dimensions: symptoms, activity and impact on daily life. To determine the outcome, a score ranging from 1 to 100 was calculated for each individual domain and for the total score, and smaller scores indicate better health status. For this outcome measure, the symptoms component score was reported.
Time Frame: Baseline and end of treatment (Week 44/46)
Population: FAS with participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Placebo 28 Days on/Off (Placebo 28) | Placebo 14 Days on/Off (Placebo 14)
Number analyzed (Participants) | 115 | 101 | 46 | 45
Score on a scale | -8.17 (22.92) | -7.20 (20.41) | -4.23 (19.55) | 2.78 (16.16)

6. Secondary Outcome: Percentage of Participants With Occurrence of New Pathogens Present at End of Treatment (Week 44/46)
Description: New pathogens were any of the pre-specified organisms not cultured before start of study medication. There was no imputation for participants who discontinued the study prematurely.
Time Frame: End of treatment (Week 44/46)
Population: Full analysis set (FAS) included participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Number analyzed (Participants) | 141 | 137 | 138
Percentage of Participants
  No | 60.3 | 49.6 | 42.8
  Yes | 3.5 | 5.1 | 8.0

7. Secondary Outcome: Mean Change From Baseline in Patient Reported Outcome Quality of Life Questionnaire for Bronchiectasis (QoL-B) Respiratory Symptoms Domain Score at End of Treatment (Week 44/46)
Description: The QoL-B was a disease-specific questionnaire developed for non-Cystic fibrosis Bronchiectasis. It covers 8 dimensions: physical functioning, role functioning, emotional functioning, social functioning, vitality, treatment burden, health perceptions, and respiratory symptoms. Each dimension was scored separately on a scale of 0 to 100, and higher scores represent better outcomes. For this outcome measure, the respiratory symptoms domain score was reported.
Time Frame: Baseline and end of treatment (Week 44/46)
Population: FAS with participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Placebo 28 Days on/Off (Placebo 28) | Placebo 14 Days on/Off (Placebo 14)
Number analyzed (Participants) | 110 | 95 | 46 | 44
Score on a scale | 7.70 (18.50) | 6.72 (17.90) | 8.22 (16.74) | 4.45 (17.78)

8. Secondary Outcome: Mean Change From Baseline in Forced Expiratory Volume in One Second (FEV1) at End of Treatment (Week 44/46)
Description: FEV1 was defined as the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration, expressed in liters at body temperature and ambient pressure saturated with water vapor (BTPS).
Time Frame: Baseline and end of treatment (Week 44/46)
Population: FAS with participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Placebo 28 Days on/Off (Placebo 28) | Placebo 14 Days on/Off (Placebo 14)
Number analyzed (Participants) | 112 | 98 | 45 | 41
Liter | -0.012 (0.149) | -0.026 (0.226) | 0.024 (0.344) | 0.022 (0.352)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 30 days after the last study drug administration.
Groups:
- Ciprofloxacin DPI 28 Days on/Off (Cipro 28): Participants received ciprofloxacin (BAYQ3939) 32.5 mg corresponding to 50 mg DPI administered BID (every 12 hours); a treatment cycle consisted of a 28-day on-treatment phase followed by a 28-day off-treatment phase (48 weeks treatment phase = 6 active cycles).
- Pooled Placebo: Participants received matching placebo matched to ciprofloxacin 32.5 mg powder (containing 40 mg dry powder) administered BID (every 12 hours); a treatment cycle consisted of either a 28-day days on-treatment phase followed by 28-day off-treatment phase or 14-day on-treatment phase followed by 14-day off treatment phase (48 weeks treatment phase = 6 cycles and 12 cycles, respectively).
Arm/Group | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) | Pooled Placebo
Serious Adverse Events (participants affected / at risk) | 29/141 | 23/136 | 32/137
Other Adverse Events (participants affected / at risk) | 74/141 | 83/136 | 62/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) (N=141) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) (N=136) | Pooled Placebo (N=137)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal vasculitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Strangulated hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pathogen resistance (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 4 (4) | 5 (5)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Complications of transplant surgery (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urethral stricture traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 8 (9) | 17 (19)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pyometra (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciprofloxacin DPI 28 Days on/Off (Cipro 28) (N=141) | Ciprofloxacin DPI 14 Days on/Off (Cipro 14) (N=136) | Pooled Placebo (N=137)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 9 (11) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (5) | 10 (11) | 7 (7)
Chest pain (General disorders) | 5 (5) | 7 (8) | 7 (7)
Fatigue (General disorders) | 6 (6) | 12 (14) | 3 (3)
Nasopharyngitis (Infections and infestations) | 15 (20) | 16 (21) | 10 (15)
Sinusitis (Infections and infestations) | 4 (5) | 10 (12) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 9 (9) | 10 (13)
Aspergillus test positive (Investigations) | 6 (6) | 7 (8) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 9 (10) | 6 (6)
Dizziness (Nervous system disorders) | 2 (2) | 7 (7) | 1 (1)
Headache (Nervous system disorders) | 11 (14) | 14 (16) | 4 (6)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (13) | 10 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 13 (18) | 9 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (21) | 16 (26) | 9 (11)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 15 (34) | 16 (32) | 8 (10)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 6 (8) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bayer acknowledges and accepts the interest in the noncommercial scientific publication of Results. In a multicenter study the PIs will not make any publication of the results before the first multi-center publication. Proposed publication/presentation shall be provided to Bayer at least 60 days prior to the intended submission or presentation of the publication in order to allow Bayer to review it. Any difference of opinion shall be discussed.